CLINICAL TRIAL: NCT03635762
Title: DESIGN CF: Developing e-Health Systems to Improve Growth and Nutrition in CF Phase 2
Brief Title: Developing e-Health Systems to Improve Growth and Nutrition in CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Johns Hopkins University (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Gregory Sawicki, Co-Chair of Success with Therapies Research Consortium, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-P00028680; STRC- 117-18-02 (Other: Success with Therapies Research Consortium)
Record Dates: First submitted 2018-07-18; First posted 2018-08-17 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Cystic Fibrosis in Children
Keywords: Nutrition; Behavioral Intervention
MeSH Terms: interventions — Fees and Charges

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Be In Charge (Experimental): behavioral + nutrition education program
  Interventions: Behavioral: Be In Charge

INTERVENTIONS:
Behavioral: Be In Charge — comparison of pre and post-program weight and calorie intake

SUMMARY:
Being at or above the 50th percentile body mass index (BMI) for age and gender in children with cystic fibrosis (CF) is associated with better lung functioning as measured by FEV1, yet diet is one of the least adhered to components of the CF treatment regimen. Investigators at Cincinnati Children's Hospital Medical Center (CCHMC) have developed an efficacious behavioral plus nutrition education program (Be In Charge) that improves adherence to dietary recommendations, and promotes weight gain in children with CF.

To make Be In Charge (BIC) widely available to families of children with CF ages 3 to 10 years, the investigators translated the face-to-face intervention into a 10-week, web-based intervention (BeInCharge.org). The investigators tested it in a pilot study and the results were promising. In the first phase of the current study, the investigators worked with a team of clinicians, parents and technology developers to extend the usability and functionality of the web intervention, enable parent-clinician collaboration, and support concurrent use across multiple clinical sites. The long term goal of this research is to make BeInCharge.org available through CF Centers across the country to patients that would benefit in order to improve dietary adherence.

The current phase of this protocol is a prospective, multicenter, nonrandomized study enrolling up to 150 parents of children with CF. Participants will complete the Be In Charge program outside of CF clinic on their own time. CF Center clinicians will be able to follow the participant's progress via the Be In Charge clinician dashboard. CF center clinicians will be asked to support participating families in completing the program as clinically appropriate.

The primary study objective is to:

1. Demonstrate preliminary effectiveness on weight and calorie intake outcomes when the Be In Charge program is integrated into clinical care with implementation support for care teams.

The secondary study objectives are to:

1. Develop a well-defined, tested set of implementation strategies consolidated into a change package and an optimized technology platform that will support a dissemination trial for spreading the Be In Charge program across CF Centers.
2. Demonstrate that it is feasible and acceptable to use the Be In Charge program in clinical care and with fidelity to intervention parameters.
3. Demonstrate sustainability of the Be In Charge program through effective use by participants and clinicians.

ELIGIBILITY:
Inclusion Criteria:

The child with CF should:

1. Have documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype or one or more of the following criteria:

   1. Sweat chloride equal to or greater than 60 milliequivalents per liter (mEq/L) by quantitative pilocarpine iontophoresis test (QPIT)
   2. two well-characterized mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene
2. Be between the ages of 3 - 10 years at the time of enrollment
3. Be below the 50th percentile BMI and/or would benefit from behavioral strategies to address mealtime behaviors/have a history of struggling with recommended nutritional intake as determined by the physician, dietitian , psychologist, or other CF Care team member

   The parent or legal authorized representative should:
4. Have regular access to a desktop device with internet or an iOS or Android mobile device with internet (tablet with internet or smartphone with a data plan)
5. Be a primary caregiver who is routinely involved in and has primary responsibility for mealtimes with their child
6. Be willing to use Be in Charge and have clinical care team review progress

Exclusion Criteria:

The child with CF should not:

1. Have a medical condition that would affect diet or growth (e.g., CF related diabetes)
2. Be receiving parenteral nutrition or nutritional supplements via a feeding tube (e.g G-tube, J-tube, nasogastric tube) at time of enrollment
3. Have a significant developmental disability/delay
4. Have a sputum culture positive for Burkholderia Cepacia
5. Have a forced expiratory volume in the first second of expiration (FEV1) of less than 40% Predicted if the child is able to reliably perform spirometry according to American Thoracic Society (ATS) guidelines.

   Parents/legal authorized representatives will be excluded if they:
6. Are unable to speak or read English.
7. Have a major psychiatric disorder or disability that would interfere with their ability to use the program or participate in the study.
8. Participated in Phase I of the DESIGN CF study.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in weight pre- to post-treatment | Baseline and Post-Treatment Assessment (approx. Week 10)
  Weight measured in kilograms in CF Clinic at beginning and end of treatment program
Change in caloric intake pre- to post-treatment | Completion of BeInCharge.org Module 1 (approx. week 1) and Completion of BeInCharge.org Module 7 (approx. week 7)
  Parent-reported average daily caloric intake calculated from food and beverages entered into study diet tracking mobile application between modules 1-2 and modules 6-7 of program

SECONDARY OUTCOMES:
Change in percentage of the Estimate Energy Requirement pre- to post-treatment | Completion of BeInCharge.org Module 1 (approx. week 1) and Completion of BeInCharge.org Module 7 (approx. week 7)
  Average percentage of Estimated Energy Requirement consumed per day at beginning and end of treatment calculated using age, gender, activity level and parent-reported daily caloric intake data from food and beverage entered into study diet tracking mobile application between modules 1-2 and modules 6-7 of program
Change in Body Mass Index z-score pre- to post-treatment | Baseline and Post-Treatment Assessment (approx. Week 10)
  Body Mass Index z-scores calculated from weight, height, age and gender based on Center for Disease Control growth charts
Percent eligible participants with access to technology | up to day 1
  Participant self-report of regular access to a desktop device with internet or an iOS or Android mobile device with internet (tablet with internet or smartphone with a data plan)
Percent eligible participants who agree to use the BeInCharge program | up to day 1
  Based on participant enrollment in study
Average number of minutes for clinicians to introduce Be In Charge program to participant | Baseline
  Clinician self-report of time spent during clinic visit introducing the BeInCharge program and discussing its use in the patient's care, collected at end of baseline clinic visit
Percent of participants that begin registration for BeInCharge.org program | Start of BeInCharge.org registration (approx. 1 day)
  Collected from BeInCharge.org platform user metrics and based on date of enrollment and date of completion of first screen of program (set password screen)
Percent of participants who complete registration for BeInCharge.org program | Completion of BeInCharge.org registration (approx. 1 day)
  Collected from BeinCharge.org platform user metrics and based on date of enrollment and date of completion of last program registration screen (tutorials screen)
Percent of participants who complete BeInCharge.org program | Completion of BeInCharge.org (approx. week 7)
  Collected from BeInCharge.org platform user metrics and based on completion of final screen of final module (module 7, congratulations screen)
BeInCharge.org program Ease of Use for clinicians assessed by Likert scale | Post-Treatment (approx. Week 10)
  Clinician single-item self-report to the question, "How easy was it to use BIC.org with [patient name]?" assessed by 5-point Likert scale. Values range from 1-5 with higher values indicating greater ease of use. Collected at the end of the program for each patient.
Clinician satisfaction with using the BeInCharge.org program with each specific patient assessed by Likert scale | Post-Treatment (approx. Week 10)
  Clinician single-item self-report to the question "How satisfied were you with using BIC.org with [patient name]? assessed by 5-point Likert scale. Values range from 1-5 with higher values indicating greater satisfaction. Collected at the end of the program for each patient.
Participant satisfaction with using the BeInCharge.org program assessed by Likert scale | Post-Treatment (approx. Week 10)
  Participant single-item self-report to the question "How satisfied were you with BIC.org?" assessed by 5-point Likert scale. Values range from 1-5 with higher values indicating greater satisfaction. Collected at the end of the program for each participant.

OTHER OUTCOMES:
Percent of participants that finish BeInCharge.org program registration on the same day as started | Completion of BeInCharge.org registration (approx. 1 day)
  Collected from BeInCharge.org user metrics and based on dates of participant completion of first and last registration screens
Average number of days between completing BeInCharge.org program registration and starting first program module | Start of BeInCharge.org Module 1 (approx. 1 week)
  Collected from BeInCharge.org user metrics and based on dates of participant completion of registration screen (tutorials screen) and start of module 1 (overview screen)
Percent of participants that complete first program module within 1 week | Completion of BeInCharge.org Module 1 (approx. 1 week)
  Collected from BeInCharge.org user metrics and based on dates of participant actions of completing module 1 start (overview screen) and module 1 end (scheduling screen)
Percent of participants that complete first program module within 1 day | Completion of BeInCharge.org Module 1 (approx. 1 day)
  Collected from BeInCharge.org user metrics and based on dates of participant actions of completing module 1 start (overview screen) and module 1 end (scheduling screen)
Average number of BeInCharge.org program modules completed within 28 days of registration | BeInCharge.org registration completion to Day 28
  Collected from BeInCharge.org user metrics and based on dates of completion for registration and program modules
Average number of days to complete BeInCharge.org program | Completion of BeInCharge.org Module (approx. week 7)
  Collected from BeInCharge.org user metrics and based on dates of participant actions of starting module 1 and completing module 7
Percent of days with entries in the study food tracking mobile application | Start of BeInCharge.org Module 7 (approx. week 7)
  Collected from BeInCharge.org user metrics and based on a count of the number of days for which a food or beverage was entered in the food tracking mobile application from the start of module 1 to the start of module 7
Percent of participants that start program module 2 within 10 days of completing module 1 | Start of BeInCharge.org Module 2 (approx. weeks 2-3)
  Collected from BeInCharge.org user metrics and based on dates of completing module 1 and starting module 2
Percent of patients for whom a clinician reports reviewing BeInCharge.org program data prior to or during post-program visit | Post-Treatment Assessment (approx. week 10)
  Clinician self-report to a multiple choice question assessing their actions regarding platform data review for their patient collected as part of post-program assessment
3. Percent of clinicians that login to the Be In Charge Clinician dashboard weekly | Post-Treatment Assessment (approx. week 10)
  Collected from BeInCharge.org clinician dashboard metrics and based on dates of patient registration in program and dates of clinician activity on the platform

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Opipari, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (7):
- United States (7):
  - Lucile Packard Children's Hospital Stanford, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Boston Childrens Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Texas- Southwestern, Dallas, Texas
  - Children's Hospital of Richmond at VCU, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No